CLINICAL TRIAL: NCT00440193
Title: Oral Direct Factor Xa Inhibitor Rivaroxaban in Patients With Acute Symptomatic Deep-Vein Thrombosis or Pulmonary Embolism
Brief Title: Oral Direct Factor Xa Inhibitor Rivaroxaban in Patients With Acute Symptomatic Deep Vein Thrombosis - The EINSTEIN DVT Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11702a; 2006-004495-13 (EudraCT Number); 11702b (Other: Company internal)
Record Dates: First submitted 2007-02-23; First posted 2007-02-26 (Estimated); Results first posted 2013-01-24 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-01

CONDITIONS: Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban (Xarelto, BAY59-7939) (Experimental): Participants were to receive rivaroxaban 15 mg oral tablet twice daily for 3 weeks, followed by 20 mg once daily
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Enoxaparin/VKA (Active Comparator): Participants were to receive 1.0 mg/kg enoxaparin twice daily (subcutaneous) for at least 5 days, plus vitamin K antagonist (VKA) (oral) at individually titrated doses to achieve a target international normalized ratio (INR) of 2.5 (range: 2.0 to 3.0)
  Interventions: Drug: Enoxaparin followed by VKA

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — During the first 3 weeks patients will receive 15 mg rivaroxaban twice-daily. Thereafter, patients will receive rivaroxaban 20 mg once-daily. Rivaroxaban will be administered orally and should be taken with food.
  Arms: Rivaroxaban (Xarelto, BAY59-7939)
Drug: Enoxaparin followed by VKA — Enoxaparin 1.0 mg/kg twice daily with a minimal duration of 5 days. This 5 days treatment could include the period up to 36 h before randomization if enoxaparin twice-daily was used. VKA should be started as soon as possible but not later than 48 hours after randomization.
  Arms: Enoxaparin/VKA

SUMMARY:
This is a multicenter, randomized, open-label, assessor-blind, event-driven, non-inferiority program for efficacy with a study treatment duration of 3, 6 or 12 months in patients with confirmed acute symptomatic DVT without symptomatic PE (Einstein-DVT).

DETAILED DESCRIPTION:
Within the US 'Johnson & Johnson Pharmaceutical Research & Development, L.L.C.' is sponsor.

The treatment period was followed by an observational period of 30 days starting the day after the last intake of study medication, regardless of the actual duration of study drug administration. Participants who did not complete the treatment period also entered the observational period. It was also possible that participants did not enter the observational period, e.g. due to withdrawal of consent or termination of study participation. Participants who were transferring from study 11702 DVT (NCT00440193) to the extension study 11899 (NCT00439725) did not enter the observational period.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed acute symptomatic proximal DVT without symptomatic PE

Exclusion Criteria:

* Legal lower age limitations (country specific)
* Thrombectomy, insertion of a caval filter, or use of a fibrinolytic agent to treat the current episode of DVT and/or PE
* Other indication for VKA than DVT and/or PE
* The pre-randomization anti-coagulant treatment (Criteria # 4) has been prolonged from 36 hours to a maximum of 48 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3449 (Actual)
Dates: Start 2007-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (266):
- United States (21):
  - Little Rock, Arkansas
  - Redlands, California
  - Bay Pines, Florida
  - Miami, Florida
  - Idaho Falls, Idaho
  - Covington, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Albuquerque, New Mexico
  - Chapel Hill, North Carolina
  - Greensboro, North Carolina
  - Oklahoma City, Oklahoma
  - Camp Hill, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Corsicana, Texas
  - San Antonio, Texas
  - Murray, Utah
  - Salt Lake City, Utah
  - Fredericksburg, Virginia
  - Spokane, Washington
  - Tacoma, Washington
- Australia (19):
  - Garran, Australian Capital Territory
  - Darlinghurst, New South Wales
  - Gosford, New South Wales
  - Kogarah, New South Wales
  - Lismore, New South Wales
  - St Leonards, New South Wales
  - Sydney, New South Wales
  - Brisbane, Queensland
  - Redcliffe, Queensland
  - Southport, Queensland
  - Woolloongabba, Queensland
  - Adelaide, South Australia
  - Woodville South, South Australia
  - Box Hill, Victoria
  - Clayton, Victoria
  - Geelong, Victoria
  - Melbourne, Victoria
  - Fremantle, Western Australia
  - Perth, Western Australia
- Austria (5):
  - Graz, Styria
  - Vienna, Vienna
  - Feldkirch, Vorarlberg
  - Innsbruck
  - Salzburg
- Belgium (11):
  - Bruxelles - Brussel
  - Duffel
  - Genk
  - Ghent
  - Hasselt
  - Leuven
  - Lier
  - Liège
  - Namur
  - Yvoir
  - Zottegem
- Brazil (7):
  - Uberaba, Minas Gerais
  - Curitiba, Paraná
  - Londrina, Paraná
  - Botucatu, São Paulo
  - São Paulo, São Paulo
  - Sorocaba, São Paulo
  - Rio de Janeiro
- Canada (4):
  - Winnipeg, Manitoba
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
- China (8):
  - Guangzhou, Guangdong
  - Harbin, Heilongjiang
  - Wuhan, Hubei
  - Suzhou, Jiangsu
  - Shenyang, Liaoning
  - Hangzhou, Zhejiang
  - Beijing
  - Shanghai
- Czechia (6):
  - Karlovy Vary
  - Kladno
  - Ostrava
  - Ostrava-Poruba
  - Prague
  - Usti Nad Lebem
- Denmark (4):
  - Aarhus C
  - Brædstrup
  - Frederiksberg
  - Hellerup
- Seinäjoki, Finland
- France (34):
  - Agen
  - Amiens
  - Angers
  - Arras
  - Besançon
  - Bordeaux
  - Brest
  - Castelnau-le-Lez
  - Clamart
  - Clermont-Ferrand
  - Colombes
  - Créteil
  - Dijon
  - Grenoble
  - Lille
  - Limoges
  - Metz-Tessy
  - Montpellier
  - Nantes
  - Nice
  - Nîmes
  - Orthez
  - Paris
  - Pierre-Bénite
  - Roanne
  - Rouen
  - Saint-Etienne
  - Strasbourg
  - Toulon
  - Toulouse
  - Tours
  - Valenciennes
  - Vandœuvre-lès-Nancy
  - Vernon
- Germany (29):
  - Bruchsal, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Karlsbad, Baden-Wurttemberg
  - Mannheim, Baden-Wurttemberg
  - Neckargemünd, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - Augsburg, Bavaria
  - München, Bavaria
  - Würzburg, Bavaria
  - Hamburg, Hamburg
  - Darmstadt, Hesse
  - Frankfurt am Main, Hesse
  - Giessen, Hesse
  - Wiesbaden, Hesse
  - Hanover, Lower Saxony
  - Rotenburg (Wümme), Lower Saxony
  - Greifswald, Mecklenburg-Vorpommern
  - Düsseldorf, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Paderborn, North Rhine-Westphalia
  - Soest, North Rhine-Westphalia
  - Witten, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Homburg, Saarland
  - Dresden, Saxony
  - Leipzig, Saxony
  - Halle, Saxony-Anhalt
  - Magdeburg, Saxony-Anhalt
  - Berlin, State of Berlin
- Hong Kong (2):
  - Hong Kong
  - Wan Chai
- Hungary (7):
  - Budapest
  - Debrecen
  - Kecskemét
  - Kistarcsa
  - Miskolc
  - Szentes
  - Szombathely
- India (6):
  - Kochi, Kerala
  - Mumbai, Maharashtra
  - Hyderabad
  - Kolkata
  - New Delhi
  - Pune
- Indonesia (5):
  - Jakarta, Indonesia
  - Bandung
  - Jakarta
  - Medan
  - Semarang
- Israel (11):
  - Afula, Israel
  - Ashkelon, Israel
  - Beersheba, Israel
  - Haifa, Israel
  - Holon, Israel
  - Jerusalem, Israel
  - Kfar Saba, Israel
  - Petah Tikva, Israel
  - Rehovot, Israel
  - Safed, Israel
  - Tel Aviv, Israel
- Italy (13):
  - Bologna
  - Chieti
  - Cremona
  - Milan
  - Napoli
  - Padua
  - Palermo
  - Parma
  - Pavia
  - Piacenza
  - Reggio Emilia
  - Varese
  - Venezia
- Kuala Selangor, Malaysia
- Netherlands (10):
  - Amsterdam
  - Arnhem
  - Dordrecht
  - Enschede
  - Groningen
  - Hoofddorp
  - Maastricht
  - Rotterdam
  - Zwijndrecht
  - Zwolle
- New Zealand (4):
  - Auckland
  - Christchurch
  - Palmerston North
  - Wellington South
- Norway (4):
  - Fredrikstad
  - Oslo
  - Rud
  - Trondheim
- Quezon City, Philippines
- Poland (11):
  - Bialystok
  - Bydgoszcz
  - Gdansk
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Poznan
  - Torun
  - Warsaw
  - Wroclaw
- San Juan, Puerto Rico
- Singapore, Singapore
- South Africa (6):
  - Cape Town, Cape
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
  - Cape Town, Western Cape
  - Somerset West, Western Cape
  - Worcester, Western Cape
- South Korea (5):
  - Daegu, Daegu
  - Seoul, Korea
  - Daegu
  - Seoul
  - Taegu
- Spain (8):
  - Barcelona, Barcelona
  - Terrassa, Barcelona
  - Girona, Girona
  - Alcorcón, Madrid
  - Fuenlabrada, Madrid
  - Madrid, Madrid
  - Pamplona, Pamplona
  - Xàtiva, Valencia
- Sweden (5):
  - Borås
  - Gothenburg
  - Jönköping
  - Sundsvall
  - Västervik
- Switzerland (5):
  - Lausanne, Canton of Vaud
  - Zurich, Canton of Zurich
  - Genéve 14, Genève 14
  - Chur, Kanton Graubünden
  - Lucerne
- Taiwan (3):
  - Kaosiung, Kaoshiong
  - Taichung
  - Taipei
- Thailand (3):
  - Bangkok, Bangkok
  - Pathumwan, Bangkok, Thailand
  - Bangkok
- United Kingdom (5):
  - Plymouth, Devon
  - Chelmsford, Essex
  - Isleworth, Greater London
  - London, Greater London
  - London

REFERENCES:
- [Result] EINSTEIN Investigators; Bauersachs R, Berkowitz SD, Brenner B, Buller HR, Decousus H, Gallus AS, Lensing AW, Misselwitz F, Prins MH, Raskob GE, Segers A, Verhamme P, Wells P, Agnelli G, Bounameaux H, Cohen A, Davidson BL, Piovella F, Schellong S. Oral rivaroxaban for symptomatic venous thromboembolism. N Engl J Med. 2010 Dec 23;363(26):2499-510. doi: 10.1056/NEJMoa1007903. Epub 2010 Dec 3. PMID 21128814
- [Result] Cohen AT, Dobromirski M. The use of rivaroxaban for short- and long-term treatment of venous thromboembolism. Thromb Haemost. 2012 Jun;107(6):1035-43. doi: 10.1160/TH11-12-0859. Epub 2012 Feb 28. PMID 22371186
- [Result] Prins MH, Lensing AW. Derivation of the non-inferiority margin for the evaluation of direct oral anticoagulants in the treatment of venous thromboembolism. Thromb J. 2013 Jul 6;11(1):13. doi: 10.1186/1477-9560-11-13. PMID 23829521
- [Result] Prins MH, Lensing AW, Bauersachs R, van Bellen B, Bounameaux H, Brighton TA, Cohen AT, Davidson BL, Decousus H, Raskob GE, Berkowitz SD, Wells PS; EINSTEIN Investigators. Oral rivaroxaban versus standard therapy for the treatment of symptomatic venous thromboembolism: a pooled analysis of the EINSTEIN-DVT and PE randomized studies. Thromb J. 2013 Sep 20;11(1):21. doi: 10.1186/1477-9560-11-21. PMID 24053656
- [Result] Wang Y, Wang C, Chen Z, Zhang J, Liu Z, Jin B, Ying K, Liu C, Shao Y, Jing Z, Meng IL, Prins MH, Pap AF, Muller K, Lensing AW; Chinese EINSTEIN Investigators. Rivaroxaban for the treatment of symptomatic deep-vein thrombosis and pulmonary embolism in Chinese patients: a subgroup analysis of the EINSTEIN DVT and PE studies. Thromb J. 2013 Dec 16;11(1):25. doi: 10.1186/1477-9560-11-25. PMID 24341332
- [Result] Bamber L, Wang MY, Prins MH, Ciniglio C, Bauersachs R, Lensing AW, Cano SJ. Patient-reported treatment satisfaction with oral rivaroxaban versus standard therapy in the treatment of acute symptomatic deep-vein thrombosis. Thromb Haemost. 2013 Oct;110(4):732-41. doi: 10.1160/TH13-03-0243. Epub 2013 Jul 11. PMID 23846019
- [Result] van Bellen B, Bamber L, Correa de Carvalho F, Prins M, Wang M, Lensing AW. Reduction in the length of stay with rivaroxaban as a single-drug regimen for the treatment of deep vein thrombosis and pulmonary embolism. Curr Med Res Opin. 2014 May;30(5):829-37. doi: 10.1185/03007995.2013.879439. Epub 2014 Jan 22. PMID 24432872
- [Result] Cano SJ, Lamping DL, Bamber L, Smith S. The Anti-Clot Treatment Scale (ACTS) in clinical trials: cross-cultural validation in venous thromboembolism patients. Health Qual Life Outcomes. 2012 Sep 26;10:120. doi: 10.1186/1477-7525-10-120. PMID 23013426
- [Derived] Dobesh PP, Volkl AA, Pap AF, Damaraju CV, Levitan B, Yuan Z, Amin AN. Benefit-Risk Assessment of Rivaroxaban in Older Patients With Nonvalvular Atrial Fibrillation or Venous Thromboembolism. Drugs Aging. 2025 May;42(5):469-484. doi: 10.1007/s40266-025-01192-7. Epub 2025 Mar 31. PMID 40163217
- [Derived] Yang L, Wu J. Cost-effectiveness of rivaroxaban compared with enoxaparin plus warfarin for the treatment of hospitalised acute deep vein thrombosis in China. BMJ Open. 2020 Jul 30;10(7):e038433. doi: 10.1136/bmjopen-2020-038433. PMID 32737096
- [Derived] Ten Cate H, Lensing AWA, Weitz JI, Middeldorp S, Beyer-Westendorf J, Kubitza D, Brighton T, Raskob GE, Mismetti P, Prandoni P, Gebel M, Prins MH. The prothrombin time does not predict the risk of recurrent venous thromboembolism or major bleeding in rivaroxaban-treated patients. Thromb Res. 2018 Oct;170:75-83. doi: 10.1016/j.thromres.2018.08.008. Epub 2018 Aug 15. PMID 30121419
- [Derived] Di Nisio M, Vedovati MC, Riera-Mestre A, Prins MH, Mueller K, Cohen AT, Wells PS, Beyer-Westendorf J, Prandoni P, Bounameaux H, Kubitza D, Schneider J, Pisters R, Fedacko J, Fontes-Carvalho R, Lensing AW. Treatment of venous thromboembolism with rivaroxaban in relation to body weight. A sub-analysis of the EINSTEIN DVT/PE studies. Thromb Haemost. 2016 Sep 27;116(4):739-46. doi: 10.1160/TH16-02-0087. Epub 2016 Aug 18. PMID 27535349
- [Derived] Prins MH, Lensing AW, Brighton TA, Lyons RM, Rehm J, Trajanovic M, Davidson BL, Beyer-Westendorf J, Pap AF, Berkowitz SD, Cohen AT, Kovacs MJ, Wells PS, Prandoni P. Oral rivaroxaban versus enoxaparin with vitamin K antagonist for the treatment of symptomatic venous thromboembolism in patients with cancer (EINSTEIN-DVT and EINSTEIN-PE): a pooled subgroup analysis of two randomised controlled trials. Lancet Haematol. 2014 Oct;1(1):e37-46. doi: 10.1016/S2352-3026(14)70018-3. Epub 2014 Sep 28. PMID 27030066
- [Derived] Bauersachs RM, Lensing AW, Prins MH, Kubitza D, Pap AF, Decousus H, Beyer-Westendorf J, Prandoni P. Rivaroxaban versus enoxaparin/vitamin K antagonist therapy in patients with venous thromboembolism and renal impairment. Thromb J. 2014 Nov 24;12:25. doi: 10.1186/1477-9560-12-25. eCollection 2014. PMID 25750589
- [Derived] Wells PS, Gebel M, Prins MH, Davidson BL, Lensing AW. Influence of statin use on the incidence of recurrent venous thromboembolism and major bleeding in patients receiving rivaroxaban or standard anticoagulant therapy. Thromb J. 2014 Nov 26;12:26. doi: 10.1186/1477-9560-12-26. eCollection 2014. PMID 25698905

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with confirmed acute proximal symptomatic deep vein thrombosis (DVT) without symptomatic pulmonary embolism (PE) were recruited at specialized study sites.
Pre-assignment Details: Out of 3459 participants screened, 10 failed screening due to protocol violations, and 3449 participants were randomized (1731 to rivaroxaban and 1718 to enoxaparin/VKA).
Period: Treatment Period
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Started | 1731 | 1718
Participants Received Treatment | 1718 | 1711
Completed | 1426 | 1367
Not Completed | 305 | 351
Not completed — Adverse Event | 74 | 67
Not completed — Death | 19 | 22
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 12 | 18
Not completed — Physician Decision | 3 | 6
Not completed — Protocol Violation | 16 | 19
Not completed — Withdrawal by Subject | 36 | 77
Not completed — Clinical endpoint reached | 28 | 25
Not completed — Study terminated by sponsor | 102 | 94
Not completed — Protocol driven decision point | 2 | 2
Not completed — Switch to commercial drug | 0 | 2
Not completed — Technical problems | 1 | 1
Not completed — Participant convenience | 5 | 2
Not completed — Participant did not receive treatment | 7 | 13
Not completed — Site closed by investigator | 0 | 2
Period: Observational Period
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Started | 1425 (All participants who took any study medication and entered the observational period.) | 1407 (All participants who took any study medication and entered the observational period.)
Completed | 1380 | 1369
Not Completed | 45 | 38
Not completed — Adverse Event | 2 | 2
Not completed — Death | 15 | 20
Not completed — Lost to Follow-up | 12 | 8
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 11 | 8
Not completed — Physician Decision | 1 | 0
Not completed — Clinical endpoint reached | 1 | 0
Not completed — Participant convenience | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA | Total
Number analyzed (Participants) | 1731 | 1718 | 3449
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (16.4) | 56.4 (16.3) | 56.1 (16.4)
Age, Customized [Number; unit: participants]
  18 - < 40 years | 314 | 279 | 593
  40 - < 60 years | 642 | 662 | 1304
  60 - < 75 years | 530 | 519 | 1049
  ≥ 75 years | 245 | 258 | 503
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 738 | 751 | 1489
  Male | 993 | 967 | 1960

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Symptomatic Recurrent Venous Thromboembolism [VTE] (i.e. the Composite of Recurrent Deep Vein Thrombosis [DVT] or Fatal or Non-fatal Pulmonary Embolism [PE]) Until the Intended End of Study Treatment
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based on either compression ultrasound (for DVT), venography (for DVT), spiral computed tomography (CT) scanning (for PE), pulmonary angiography (for PE), ventilation/perfusion lung scan (for PE), lung scintigraphy (for PE), autopsy (for fatal PE) or unexplained death for which DVT/PE could not be ruled out (for fatal PE), and/or case summaries.
Time Frame: 3-, 6- or 12-month study treatment period
Population: The intention-to-treat (ITT) population consisted of all randomized participants with valid informed consent. Participants were analyzed according to the treatment assigned at randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 1731 | 1718
Percentage of participants | 2.1 | 3.0
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Enoxaparin/VKA; The rivaroxaban to comparator hazard ratio was computed with a 95% CI (confidence interval) (two-sided testing). Based on this model, rivaroxaban would be considered at least as effective as the comparator if the upper limit of the CI was less than 2.0; Test type: Non-Inferiority or Equivalence — Assuming equal efficacy, a total of 88 events was calculated to give a power of 90% to prove that rivaroxaban is at least as effective as the comparator, considering a non-inferiority upper CI margin for the hazard ratio of 2.0 (two-sided α=0.05). A mean incidence for the primary efficacy outcome of 3% was expected and at least 1465 participants per group were determined to be necessary. This number was to be adjusted based on the observed overall incidence of symptomatic recurrent VTE; p < 0.0001, Regression, Cox; Stratified by intend treatment duration, adjusted for presence of active malignancy at baseline; Hazard Ratio (HR) = 0.68, 95% CI [0.44 to 1.04], Standard Error of Mean 0.2179 — The standard error of the log hazard ratio was estimated

2. Secondary Outcome: Percentage of Participants With the Composite Variable Comprising Recurrent DVT, Non-fatal PE and All Cause Mortality Until the Intended End of Study Treatment
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based on either compression ultrasound (for DVT), venography (for DVT), spiral computed tomography (CT) scanning (for PE), pulmonary angiography (for PE), ventilation/perfusion lung scan (for PE), lung scintigraphy (for PE), autopsy (for deaths), results/films/images of confirmatory testing, and/or case summaries.
Time Frame: 3-, 6- or 12-month study treatment period
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 1731 | 1718
Percentage of participants | 4.0 | 5.1
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Enoxaparin/VKA; Test type: Superiority or Other; p = 0.044, Regression, Cox — Nominal p-value; Stratified by intend treatment duration, adjusted for presence of active malignancy at baseline; Hazard Ratio (HR) = 0.72, 95% CI [0.53 to 0.99], Standard Error of Mean 0.1616 — The standard error of the log hazard ratio was estimated

3. Secondary Outcome: Percentage of Participants With an Event for Net Clinical Benefit 1 Until the Intended End of Study Treatment
Description: Net clinical benefit 1: composite of recurrent DVT or non-fatal or fatal PE, and major bleeding. Major bleeding was overt bleeding associated with 2 g/dL or greater fall in hemoglobin, leading to a transfusion of ≥2 units, occurring in a critical site or contributing to death. Net clinical benefit was considered greater in those participants with fewer composite events. All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment, based on either compression ultrasound, venography, spiral computed tomography scanning, pulmonary angiography, ventilation/perfusion lung scan, lung scintigraphy, autopsy or unexplained death for which DVT/PE could not be ruled out, results/films/images of confirmatory testing, and/or case summaries.
Time Frame: 3-, 6- or 12-month study treatment period
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 1731 | 1718
Percentage of participants | 2.9 | 4.2
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Enoxaparin/VKA; Test type: Superiority or Other; p = 0.027, Regression, Cox — Nominal p-value; Stratified by intend treatment duration, adjusted for presence of active malignancy at baseline; Hazard Ratio (HR) = 0.67, 95% CI [0.47 to 0.95], Standard Error of Mean 0.1828 — The standard error of the log hazard ratio was estimated

4. Secondary Outcome: Percentage of Participants With Recurrent DVT Until the Intended End of Study Treatment
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based on either compression ultrasound, venography, results/films/images of confirmatory testing, and/or case summaries.
Time Frame: 3-, 6- or 12-month study treatment period
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 1731 | 1718
Percentage of participants | 0.9 | 1.6

5. Secondary Outcome: Percentage of Participants With Clinically Relevant Bleeding, Treatment-emergent (Time Window: Until 2 Days After Last Dose)
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Clinically relevant bleeding included major bleeding (overt bleeding associated with 2 g/dL or greater fall in hemoglobin, leading to a transfusion of 2 or more units of packed red blood cells or whole blood, occurring in a critical site or contributing to death) and non-major bleeding associated with medical intervention, unscheduled physician contact, (temporary) cessation of study treatment, discomfort for the participants such as pain, or impairment of activities of daily life.
Time Frame: 3-, 6- or 12-month study treatment period
Population: The valid-for-safety analysis population consisted of all participants who were randomized with valid informed consent and received at least one dose of anticoagulant study treatment after randomization (i.e. enoxaparin, warfarin, acenocoumarol, rivaroxaban). Participants were analyzed according to the treatment they actually received.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 1718 | 1711
Percentage of participants | 8.1 | 8.1
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Enoxaparin/VKA; Test type: Superiority or Other; p = 0.77, Regression, Cox — Nominal p-value; Stratified by intend treatment duration, adjusted for presence of active malignancy at baseline; Hazard Ratio (HR) = 0.97, 95% CI [0.76 to 1.22], Standard Error of Mean 0.1204 — The standard error of the log hazard ratio was estimated

6. Secondary Outcome: Percentage of Participants With All Deaths
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based on either autopsy, results/films/images of confirmatory testing, and/or case summaries.
Time Frame: 3-, 6- or 12-month study treatment period
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 1718 | 1711
Percentage of participants
  All post-randomization | 2.4 | 3.0
  Treatment-emergent (time window: 2 days) | 1.0 | 1.1
  Treatment-emergent (time window: 7 days) | 1.2 | 1.5

7. Secondary Outcome: Percentage of Participants With Other Vascular Events, On-treatment (Time Window: Until 1 Day After Last Dose)
Description: All pre-defined vascular events (ST segment elevation myocardial infarction, non ST segment elevation myocardial infarction, unstable angina, ischemic stroke, transient ischemic attack, non-central nervous system systemic embolism or vascular death) were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based results/films/images of confirmatory testing, and/or case summaries.
Time Frame: 3-, 6- or 12-month study treatment period
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 1718 | 1711
Percentage of participants | 0.7 | 0.8

8. Other Pre Specified Outcome: Percentage of Participants With the Individual Components of Efficacy Outcomes Until the Intended End of Study Treatment
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment, based on either compression ultrasound, venography, spiral computed tomography scanning, pulmonary angiography, ventilation/perfusion lung scan, lung scintigraphy, autopsy or unexplained death for which DVT/PE could not be ruled out, results/films/images of confirmatory testing, and/or case summaries. Major bleeding was overt bleeding associated with 2 g/dL or greater fall in hemoglobin, leading to a transfusion of ≥2 units, occurring in a critical site or contributing to death.
Time Frame: 3-, 6- or 12-month study treatment period
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 1731 | 1718
Percentage of participants
  Death (PE) | 0.06 | 0
  Death (PE cannot be excluded) | 0.2 | 0.3
  Symptomatic PE and DVT | 0.06 | 0
  Symptomatic recurrent PE only | 1.2 | 1.0
  Symptomatic recurrent DVT only | 0.8 | 1.6
  Death (bleeding) | 0.06 | 0.3
  Death (cardiovascular) | 0.1 | 0.2
  Death (other) | 1.8 | 2.0
  Major bleeding | 0.9 | 1.3

9. Other Pre Specified Outcome: Percentage of Participants With Symptomatic Recurrent Venous Thromboembolism [VTE] (i.e. the Composite of Recurrent Deep Vein Thrombosis [DVT] or Fatal or Non-fatal Pulmonary Embolism [PE]) During Observational Period
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based on either compression ultrasound (for DVT), venography (for DVT), spiral computed tomography (CT) scanning (for PE), pulmonary angiography (for PE), ventilation/perfusion lung scan (for PE), lung scintigraphy (for PE), autopsy (for fatal PE) or unexplained death for which DVT/PE could not be ruled out (for fatal PE), results/films/images of confirmatory testing, and/or case summaries.
Time Frame: Up to 30 days after the last intake of study medication
Population: Participants entering the observational period were participants for whom the investigator indicated on the eCRF (electronic case report form) that the participant entered the observational period or had a confirmed event more than one day and up to 30 days after the last dose as a component of the respective composite outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 1425 | 1408
Percentage of participants | 0.8 | 0.5

10. Other Pre Specified Outcome: Percentage of Participants With the Composite Variable Comprising Recurrent DVT, Non-fatal PE and All Cause Mortality During Observational Period
Description: as for outcome 2
Time Frame: Up to 30 days after the last intake of study medication
Population: Participants entering the observational period were participants for whom the investigator indicated on the eCRF that the participant entered the observational period or had a confirmed event more than one day and up to 30 days after the last dose as a component of the respective composite outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 1430 | 1413
Percentage of participants | 2.2 | 1.8

11. Other Pre Specified Outcome: Percentage of Participants With an Event for Net Clinical Benefit 1 During Observational Period
Description: Net clinical benefit 1: composite of recurrent DVT or non-fatal or fatal PE or major bleeding. Major bleeding was overt bleeding associated with 2 g/dL or greater fall in hemoglobin, leading to a transfusion of ≥2 units, occurring in a critical site or contributing to death. Net clinical benefit was considered greater in those participants with fewer composite events. All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment, based on either compression ultrasound, venography, spiral computed tomography scanning, pulmonary angiography, ventilation/perfusion lung scan, lung scintigraphy, autopsy or unexplained death for which DVT/PE could not be ruled out, results/films/images of confirmatory testing, and/or case summaries.
Time Frame: Up to 30 days after the last intake of study medication
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 1425 | 1410
Percentage of participants | 1.1 | 1.1

12. Other Pre Specified Outcome: Percentage of Participants With Recurrent DVT During Observational Period
Description: as for outcome 4
Time Frame: Up to 30 days after the last intake of study medication
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 1425 | 1408
Percentage of participants | 0.6 | 0.3

13. Other Pre Specified Outcome: Percentage of Participants With the Individual Components of Efficacy Outcomes During Observational Period
Description: as for outcome 8
Time Frame: Up to 30 days after the last intake of study medication
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 1425 | 1408
Percentage of participants
  Death (PE) | 0 | 0
  Death (PE cannot be excluded) | 0.07 | 0.07
  Symptomatic PE and DVT | 0 | 0
  Symptomatic recurrent PE only | 0.3 | 0.1
  Symptomatic recurrent DVT only | 0.6 | 0.3
  Death (bleeding) | 0.07 | 0.1
  Death (cardiovascular) | 0.07 | 0.3
  Death (other) | 1.3 | 0.8
  Major bleeding | 0.2 | 0.6

14. Post Hoc Outcome: Percentage of Participants With an Event for Net Clinical Benefit 2 Until the Intended End of Study Treatment
Description: Net clinical benefit 2: composite of recurrent DVT or non-fatal or fatal PE, major bleeding. Major bleeding was overt bleeding associated with 2 g/dL or greater fall in hemoglobin, leading to transfusion of ≥2 units, occurring in a critical site or contributing to death, cardiovascular death, myocardial infarction, stroke, and non CNS (central nervous system) systemic embolism. Net clinical benefit was considered greater in those participants with fewer composite events. All events confirmed by independent committee blinded to treatment, based on compression ultrasound, venography, spiral CT scan, pulmonary angiography, ventilation/perfusion lung scan, lung scintigraphy, autopsy, results/films/images of confirmatory testing and/or case summaries
Time Frame: 3-, 6- or 12-month study treatment period
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 1731 | 1718
Percentage of participants | 3.6 | 4.7

15. Post Hoc Outcome: Percentage of Participants With an Event for Net Clinical Benefit 2 During Observational Period
Description: Net clinical benefit 2: composite of recurrent DVT or non-fatal or fatal PE, major bleeding, cardiovascular death, myocardial infarctions, stroke, or non CNS systemic embolism. Major bleeding was associated with 2 g/dL or greater fall in hemoglobin, leading to a transfusion of ≥2 units, occurring in a critical site or contributing to death. Net clinical benefit was considered greater in those participants with fewer composite events. All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment, based on either compression ultrasound (DVT), venography (DVT), spiral CT scanning (PE), pulmonary angiography ( PE), ventilation/perfusion lung scan (PE), lung scintigraphy (PE), autopsy or unexplained death for which DVT/PE could not be ruled out, results/films/images of confirmatory testing, and/or case summaries.
Time Frame: Up to 30 days after the last intake of study medication
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Number analyzed (Participants) | 1426 | 1410
Percentage of participants | 1.2 | 1.3

ADVERSE EVENTS:
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin/VKA
Serious Adverse Events (participants affected / at risk) | 222/1718 | 252/1711
Other Adverse Events (participants affected / at risk) | 241/1718 | 212/1711
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (Xarelto, BAY59-7939) (N=1718) | Enoxaparin/VKA (N=1711)
Anaemia (Blood and lymphatic system disorders) | 11 | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 5 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 3
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 3
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 3
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0
Aortic valve disease (Cardiac disorders) | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 0 | 1
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Basedow's disease (Endocrine disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Blepharochalasis (Eye disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 2
Eye haemorrhage (Eye disorders) | 1 | 0
Hyphaema (Eye disorders) | 1 | 0
Maculopathy (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Vitreous detachment (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 2
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 3
Haematochezia (Gastrointestinal disorders) | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Intestinal dilatation (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 5 | 4
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1
Retroperitoneal fibrosis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 2 | 0
Abdominal wall cyst (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 0
Hernial eventration (Gastrointestinal disorders) | 0 | 1
Intestinal mass (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 3 | 1
Death (General disorders) | 2 | 1
Generalised oedema (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 1
Multi-organ failure (General disorders) | 3 | 2
Oedema peripheral (General disorders) | 3 | 0
Pelvic mass (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 2
Sudden death (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Medical device complication (General disorders) | 0 | 1
Device occlusion (General disorders) | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Hepatic mass (Hepatobiliary disorders) | 1 | 0
Liver transplant rejection (Immune system disorders) | 0 | 1
Abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 3 | 1
Cellulitis (Infections and infestations) | 3 | 4
Dengue fever (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Endocarditis staphylococcal (Infections and infestations) | 0 | 1
Epiglottitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 2
Escherichia sepsis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 4
Influenza (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 3
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Mastitis (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 10
Postoperative wound infection (Infections and infestations) | 1 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 7
Septic shock (Infections and infestations) | 1 | 4
Tracheobronchitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 5 | 3
Viral infection (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Incision site abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1
Cardiac valve vegetation (Infections and infestations) | 0 | 1
Cerebral toxoplasmosis (Infections and infestations) | 0 | 1
Infective aneurysm (Infections and infestations) | 1 | 0
Wound abscess (Infections and infestations) | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 2
Lung infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 2
Device related infection (Infections and infestations) | 0 | 1
Incision site infection (Infections and infestations) | 0 | 1
Post procedural sepsis (Infections and infestations) | 0 | 1
Accident (Injury, poisoning and procedural complications) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 2
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Induced abortion haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1
Gastrointestinal disorder postoperative (Injury, poisoning and procedural complications) | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 6
Blood bilirubin increased (Investigations) | 1 | 0
Chest X-ray abnormal (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 5
Liver function test abnormal (Investigations) | 2 | 4
Weight decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 2 | 0
Hepatic enzyme increased (Investigations) | 1 | 5
International normalised ratio fluctuation (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Tetany (Metabolism and nutrition disorders) | 1 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1
Diabetic foot (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 7
Cervix carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Large cell carcinoma of the respiratory tract stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Rectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma cutis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ear neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Penis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 2
Epilepsy (Nervous system disorders) | 1 | 1
Facial palsy (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 1
Hypoglycaemic coma (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Mononeuritis (Nervous system disorders) | 1 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 4
IIIrd nerve paresis (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 4 | 7
Parkinson's disease (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Complex regional pain syndrome (Nervous system disorders) | 0 | 1
Cerebral arteriosclerosis (Nervous system disorders) | 1 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Post abortion haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Acute psychosis (Psychiatric disorders) | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 3 | 2
Panic attack (Psychiatric disorders) | 1 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Anuria (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 4 | 8
Hydronephrosis (Renal and urinary disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 3
Menorrhagia (Reproductive system and breast disorders) | 5 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Penile swelling (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Scrotal swelling (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 | 2
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wegener's granulomatosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Scar (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Abortion induced (Surgical and medical procedures) | 0 | 1
Bladder catheter removal (Surgical and medical procedures) | 1 | 0
Uterine polypectomy (Surgical and medical procedures) | 0 | 1
Ileostomy closure (Surgical and medical procedures) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
Arterial thrombosis limb (Vascular disorders) | 1 | 1
Arteriosclerosis (Vascular disorders) | 0 | 2
Circulatory collapse (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 4
Hypertension (Vascular disorders) | 2 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 2
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Post thrombotic syndrome (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Femoral artery occlusion (Vascular disorders) | 1 | 0
Iliac artery stenosis (Vascular disorders) | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
Extremity necrosis (Vascular disorders) | 0 | 1
Arterial haemorrhage (Vascular disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 0
May-Thurner syndrome (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (Xarelto, BAY59-7939) (N=1718) | Enoxaparin/VKA (N=1711)
Nasopharyngitis (Infections and infestations) | 100 | 91
Headache (Nervous system disorders) | 91 | 70
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 90 | 74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less